CLINICAL TRIAL: NCT01297712
Title: On-Site Endoscopic Prediction of Polyp Histology During Screening Colonoscopy
Brief Title: Endoscopic Assessment of Polyp Histology
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: enrollment terminated, analysis ongoing
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Principal Investigator, Prof. Dr. Thomas Rösch, Director, Universitätsklinikum Hamburg-Eppendorf
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: iScan study-1
Record Dates: First submitted 2011-02-14; First posted 2011-02-17 (Estimated); Last update posted 2019-06-07 (Actual); Status verified 2019-04

CONDITIONS: Colonic Polyps
Keywords: screening colonoscopy; adenoma; hyperplastic polyp; differential diagnosis
MeSH Terms: conditions — Colonic Polyps; Adenoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Hi Line (Active Comparator): This arm is examined with latest generation HDTV colonoscopes
  Interventions: Device: Latest generation colonoscopy as diagnostic instrument
- Classic Line (No Intervention): control group undergoing colonoscopy with older generation scope currently in use in most centers

INTERVENTIONS:
Device: Latest generation colonoscopy as diagnostic instrument — this endoscope is used as compared to an older generations cope (classic line) currently in use
  Other Names: Hi Line colonoscopy; IScan Colonoscope
  Arms: Hi Line

SUMMARY:
Polyps found during screening colonoscopy have to be removed or at least biopsied. Attempts to save costs include endoscopic assessment of polyps with regards to differential diagnoses between adenomas (which have to be removed) and hyperplastic polyps (could be left in place or removed and not examined histologically). Such a concept would only be feasible if endoscopy can make the differential diagnosis with high accuracy. Such high accuracy rates - between 80% and 95% - have been reported from reference centers with specific scientific interest. The investigators want to test whether these results a) can be reproduced in the private practice setting performing large-volume screening colonoscopies and b) whether latest generation endoscopes provide benefit in terms of better accuracy.

DETAILED DESCRIPTION:
Patients undergoing screening colonoscopy will be randomized to the use of two different colonoscopes, namely the latest generation (Pentax iScan, Hi Line) versus the previous generation (Classic Line). On withdrawal, all polyps found will be diagnosed according to their pit pattern (classification scheme mit example images provided) and a differential diagnosis made during the live examination. Pit patterns I/II will be classified as hyperplastic polyps, patterns III-V as adenomas (in a subgroup IV and V will be classified as pre-/malignant). All polyps will be photographed from near distance to allow for later blinded review which will be done on patients with only one polyp (to avoid mix-up of polyps) by 3 examiners and 2 independent hospital experts.

ELIGIBILITY:
Inclusion Criteria:

* All patients undergoing screening colonoscopy

Exclusion Criteria:

* Missing consent
* No screening colonoscopy (diagnostic colonoscopy because of symptoms)

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1069 (Actual)
Dates: Start 2009-09; Primary Completion 2010-11 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Accuracy (sensitivity/specificity) of HDTV/iScan image technology (Hi Line) versus conventional colonoscopy (classic Line) in the diagnosis of adenomas versus hyperplastic polyps | 14 months

SECONDARY OUTCOMES:
Comparison of online accuracy during colonoscopy with later blinded image assessment in the differential diagnosis of adenomas versus hyperplastic polyps | 14 months

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Rösch, MD, Principal Investigator — Universitätsklinikum Hamburg-Eppendorf
Locations (1):
- University Hospital Hamburg-Eppendorf, Hamburg, Germany

REFERENCES:
- [Result] Schachschal G, Mayr M, Treszl A, Balzer K, Wegscheider K, Aschenbeck J, Aminalai A, Drossel R, Schroder A, Scheel M, Bothe CH, Bruhn JP, Burmeister W, Stange G, Bahr C, Kiesslich R, Rosch T. Endoscopic versus histological characterisation of polyps during screening colonoscopy. Gut. 2014 Mar;63(3):458-65. doi: 10.1136/gutjnl-2013-304562. Epub 2013 Jun 28. PMID 23812324